CLINICAL TRIAL: NCT05984407
Title: EFFECTS OF EXTRACORPOREAL CYTOKINE ELIMINATION ON HEMODYNAMIA AND MORTALITY IN CRITICAL PATIENTS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hakan Küçükkepeci (Other)
Responsible Party: Sponsor-Investigator, Hakan Küçükkepeci, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Organization: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Other Study IDs: 652779
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Cytokine Hemadsorption Therapy in Critically Ill Patients Who Have no Microbiological Findings and Develop Vasoplegic Shock
Keywords: vasoplegic shock, cytokine hemadsorption, hemodynamics, mortality, cytokine storm
MeSH Terms: conditions — Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with vasoplegic shock: Application of cytokine hemadsorption therapy in patients with vasoplegic shock without microbiological findings
  Interventions: Procedure: cytokine hemadsorption therapy

INTERVENTIONS:
Procedure: cytokine hemadsorption therapy — Observation of cytokine hemadsorption therapy in critically ill patients who have no microbiological findings and develop vasoplegic shock.

SUMMARY:
Observation of the effects of cytokine adsorbent hemadsorption therapy on hemodynamics and mortality in critically ill patients who developed vasoplegic shock due to hyperinflammation without microbiological findings in the intensive care unit.

DETAILED DESCRIPTION:
Observation of the effects of cytokine adsorbent hemadsorption therapy on hemodynamics and mortality in critically ill patients who developed vasoplegic shock due to hyperinflammation without microbiological findings and met the inclusion criteria in the Intensive Care Unit between 01.08.2023 and 01.02.2024

ELIGIBILITY:
Inclusion Criteria:

* C-reactive protein (CRP) ≥ 100 mg/l
* Procalcitonin (PCT) < 2 ng/l
* Patients aged 18-80 years who were treated with cytokine adsorption due to vasoplegic shock

Exclusion Criteria:

* Patients under 18 years of age
* Patients with suspected or proven bacterial cause of vasoplegic shock.
* Those who did not approve to participate in the study
* Patients without vasoplegic shock
* Patients with CRP < 100 mg/l, PCT ≥ 2 μg/L

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty patients who met the inclusion criteria were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
The time to resolution of vasoplegic shock within days. | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
7-day mortality | 7 days
mortality until discharge from hospital | From enrollment to the end of treatment at 12 weeks
Interleukin 1 beta level on day 1 | one day
Interleukin 10 level on day 1 | one day
Interleukin 6 level on day 1 | one day
TNF - α level on day 1 | one day
Interleukin 1 beta level on day 3 | 3 days
Interleukin 10 level on day 3 | 3 days
Interleukin 6 level on day 3 | 3 days
TNF - α level on day 3 | 3 days
mechanical ventilation need and duration | From enrollment to the end of treatment at 12 weeks
duration of treatment in the intensive care unit | From enrollment to the end of treatment at 12 weeks
dose of catecholamine | From enrollment to the end of treatment at 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşcıoğlu City Hospital, Istanbul, Şişli, Turkey (Türkiye)